CLINICAL TRIAL: NCT04904861
Title: Group Videoconferencing Intervention to Improve Maternal Sensitivity in Mother-infant Dyads in Primary Care in Chile : Randomized Controlled Feasibility Trial
Brief Title: Group Videoconferencing Intervention to Improve Maternal Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INTERDISCIPLINA II20029
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Parent-Child Relations; Parenting
Keywords: maternal sensitivity; videoconferencing; group intervention; primary care; telehealth
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videoconference Intervention group (Experimental): Brief group videoconferencing attachment-based intervention (sessions once a week for 4 weeks)
  Interventions: Behavioral: Videoconference intervention group
- Control group (Active Comparator): Psycho-educational intervention : They will receive brochures with information on parenting (once a week for 4 weeks)
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Videoconference intervention group — A short face-to-face dyadic group workshop focused on increasing maternal sensitivity was adapted to be carried out virtually by videoconference. The intervention considers 4 sessions, with a weekly frequency, with a minimum of 3 and a maximum of 6 dyads per group led by a monitor (psychologist). The activities are protocolized in a manual and are designed to be carried out by the mother with the baby under one year of age. .
  Arms: Videoconference Intervention group
Other: Control group — Psycho-educational intervention : They will receive brochures with information on parenting (once a week for 4 weeks) in addition to the usual care in their primary care center
  Arms: Control group

SUMMARY:
Background: Early childhood development is highly dependent on the sensitive care provided by their caregivers . Interventions focused on supporting parents to improve their sensitivity have been shown to be effective . The COVID-19 pandemic has had a great impact on mental health , with pregnant women and mothers of children under one year of age being an especially vulnerable group . On the other hand, access to mental health interventions in person is restricted by confinement measures , especially group interventions, so it is relevant to have remote interventions that support this group of mothers.

Objectives: to evaluate the feasibility and acceptability of a group videoconferencing intervention to improve maternal sensitivity aimed at mother / infant dyads attended in Primary Health Care in Chile Methodology: a randomized pilot feasibility study will be carried out with a mixed design with quantitative and qualitative evaluations. A face-to-face group intervention with proven effectiveness will be adapted to videoconferencing format , then 50 dyads will be randomized in a 3: 2 ratio to receive the videoconferencing intervention ( n=30) or the delivery of educational brochures (n=20) . The feasibility and acceptability will be evaluated assessing the participation, adherence and satisfaction in a quantitative way, in addition the qualitative evaluation will be carried out through interviews and focus groups. Changes in clinical outcomes will also be evaluated: maternal sensitivity, depressive symptoms, postnatal maternal attachment and infant socio-emotional development. This pilot study will allow the identification of the key parameters for the implementation and evaluation of the intervention, which will allow the design of an effectiveness study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a baby between 4 months and a year
* Attended at one of the participating primary care health centers
* Older than 18 years-old
* Handling Spanish fluently
* Have an electronic device that allows videoconferencing (computer, tablet or smart cell phone)

Exclusion Criteria:

* Mother with severe intellectual deficit or psychotic symptoms
* Participate in another early intervention at the health care center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention: eligibility rates | Through study completion, approximately 18 months
  percentage of eligible population that is recruitable: meets inclusion and not exclusion criteria
Feasibility of the intervention: attrition rates | Through study completion, approximately 18 months
  Attrition and follow-up rates by treatment condition.
Feasibility of the intervention: recruitment rates | Through study completion, approximately 18 months
  percentage that meets entry criteria and agrees to participate
Acceptability of the intervention : participation rates | Through study completion, approximately 18 months
  Proportion of performed sessions versus planned sessions.
Acceptability of the intervention : Satisfaction with the intervention | Through study completion, approximately 18 months
  Credibility/Expectancy Questionnaire (CEQ).Scores range from 0 to 100 with higher scores indicating higher acceptability of the intervention.
Acceptability of the intervention (qualitative assessment) | Through study completion, approximately 18 months
  Semi-structured interviews with monitors of the intervention (two psychologists) and focus groups with participating mothers (7 in total) with the aim of collecting information about the experience and identifying possible improvements

SECONDARY OUTCOMES:
Change in Maternal sensitivity | Through study completion, approximately 18 months
  Adult Sensitivity Scale (E.S.A.) rubric with 19 indicators, each indicator is scored between 1 and 3, and a higher score indicates higher sensitivity
Change in Maternal Depressive Symptoms | Through study completion, approximately 18 months
  Edinburgh Postnatal Depression Scale (EPDS). Scores range from 0 to 30, with higher scores meaning higher depressive symptomatology.
Change in Children Socio Emotional Development | Through study completion, approximately 18 months
  Ages and Stages Questionnaire (ASQ-SE). Scores range from 0 to 75 with higher scores meaning lower socio-emotional development
Change in postnatal maternal bonding | Evaluation at study entry (T0) and at the end of the intervention (T1)
  Maternal postnatal attachment scale (MPAS) : is a 19-item, self-report measure have 19 items, ranging from 1 (low bonding) to 5 (high bonding),

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - CESFAM Juan Pablo Segundo ANCORA UC Christus, Santiago
  - CESFAM Madre Teresa Calcuta ANCORA UC Christus, Santiago

REFERENCES:
- [Background] Davenport MH, Meyer S, Meah VL, Strynadka MC, Khurana R. Moms Are Not OK: COVID-19 and Maternal Mental Health. Front Glob Womens Health. 2020 Jun 19;1:1. doi: 10.3389/fgwh.2020.00001. eCollection 2020. PMID 34816146
- [Result] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Result] Britto PR, Lye SJ, Proulx K, Yousafzai AK, Matthews SG, Vaivada T, Perez-Escamilla R, Rao N, Ip P, Fernald LCH, MacMillan H, Hanson M, Wachs TD, Yao H, Yoshikawa H, Cerezo A, Leckman JF, Bhutta ZA; Early Childhood Development Interventions Review Group, for the Lancet Early Childhood Development Series Steering Committee. Nurturing care: promoting early childhood development. Lancet. 2017 Jan 7;389(10064):91-102. doi: 10.1016/S0140-6736(16)31390-3. Epub 2016 Oct 4. PMID 27717615
- [Result] Torales J, O'Higgins M, Castaldelli-Maia JM, Ventriglio A. The outbreak of COVID-19 coronavirus and its impact on global mental health. Int J Soc Psychiatry. 2020 Jun;66(4):317-320. doi: 10.1177/0020764020915212. Epub 2020 Mar 31. PMID 32233719
- [Result] Ohannessian R, Duong TA, Odone A. Global Telemedicine Implementation and Integration Within Health Systems to Fight the COVID-19 Pandemic: A Call to Action. JMIR Public Health Surveill. 2020 Apr 2;6(2):e18810. doi: 10.2196/18810. PMID 32238336
- [Derived] Binda V, Olhaberry M, Castanon C, Abarca C, Caamano C. A Group Videoconferencing Intervention (C@nnected) to Improve Maternal Sensitivity: Protocol for a Randomized Feasibility Trial. JMIR Res Protoc. 2022 Aug 15;11(8):e35881. doi: 10.2196/35881. PMID 35969451